CLINICAL TRIAL: NCT01678092
Title: Phase 1, Single Center Study Using Omalizumab in Subjects With Atopic Dermatitis
Brief Title: Single Center Study Using Omalizumab in Subjects With Atopic Dermatitis
Acronym: OXAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kari Christine Nadeau, Principle Investigator, Stanford University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 011394
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: omalizumab

SUMMARY:
A phase 1 single center study in which omalizumab is dosed normally (according to the product insert) in subjects with atopic dermatitis.

DETAILED DESCRIPTION:
A Phase I randomized, double-blinded, placebo-controlled study of Omalizumab in subjects with severe atopic dermatitis and food allergy. Subjects were to participate for 2 years. The treatment period was a 24 week period during which subjects received Omalizumab either every 2 or 4 weeks subcutaneously (as per product insert guidelines). Subjects randomized to the placebo group received sterile water every 2 or 4 weeks subcutaneously. Previous medications were standardized at equivalent doses one month prior to the first dose. The monthly laboratory assessment for each subject included a complete blood count (CBC), serum chemistries (Chem7/AST/ALT), and IgE levels.

Safety: Adverse events and clinical status were actively monitored during study visits at weeks 4, 8, 16, 20, 24, 28, 32, and 36 (up to 3 months after last study dose) the as well as reviewed in daily diaries per NIH assessment guidelines. Assessments of platelet count (CBC), liver function (LFTs), serum chemistry panel, and serum IgE were made on a monthly basis during the treatment period (24 weeks). Serum pregnancy testing was performed at screening only as part of the inclusion/exclusion criteria.

Efficacy: Efficacy parameters included a standardized SCORAD classification system, Physician's Global Assessment (PGA) score and subject/care giver global assessment for subjects at 24 weeks compared to baseline. An assessment for food allergy was made by skin prick testing and RAST performed at baseline and during or after the last dose. Diaries were also taken to assess use of concomitant medications and food allergy symptoms. In addition, one of the secondary endpoints was to assess the durability of effect of Xolair once the treatment was discontinued. This was achieved through follow-up visits 1, 2, 3, 6, 12, and 24 months after the last treatment dose. The investigators also assessed use of concomitant medications and food allergies via daily diaries for each of these assessments.

Number of subjects planned: 20 (Omalizumab 10 and Placebo 10). Number of subjects analysed: (Omalizumab 4 and Placebo 4).

Male or female aged 4-25 years. Diagnosis of severe atopic dermatitis (meeting SCORAD criteria) with at least 6 months of documented symptoms. Also with concomitant food allergy as determined by a positive skin prick testing.

Omalizumab was supplied as a sterile, white, preservative-free, lyophilized powder contained in a single-use vial that is reconstituted with Sterile Water for Injection (SWFI), USP, and administered as a subcutaneous (SC) injection. A Xolair vial contains 202.5 mg of Omalizumab, 145.5 mg sucrose, 2.8 mg L-histidine hydrochloride mono hydrate, 1.8 mg L-histidine and 0.5 mg polysorbate 20 and is designed to deliver 150 mg of Omalizumab, in 1.2 mL after reconstitution with 1.4 mL SWFI, USP. Treatment dose was determined as outlined in the product insert.

2 year study duration (24 Weeks treatment). The reference was placebo (sterile water) given subcutaneously.

The primary efficacy variables were improvement of SCORAD, Physician's Global Assessment, and Subject/Caregiver Global Assessment scores for subjects at 24 weeks compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered for inclusion in this study based on meeting all of the following criteria:

1. Male or female, aged 4 to 25 years with weight at study entry of greater than 15 kg
2. Subjects with AD involving greater than 10% of total body surface area (BSA)
3. Subjects with AD PGA score of severe at study entry
4. Subject with SCORAD score defined as severe at study entry
5. IgE level at study entry between 50 IU/mL and 3000 IU/mL
6. Subjects with documented food allergy as determined by a positive skin prick test to the specific allergen extract, defined as a wheal of at least 0.5 the diameter of the histamine produced wheal and at least 3 mm larger than the diameter of the negative control, associated with exacerbation of atopic dermatitis
7. Men and women of reproductive potential who document use of adequate contraception during the study and for 3 months after the conclusion of treatment with study drug/placebo
8. Historical documentation of atopic dermatitis on one occasion in the patient's medical record. The patient should have 6 months or more of atopic dermatitis symptoms.
9. Women of childbearing potential who have a negative pregnancy test (urine or serum) at the time of study entry -

Exclusion Criteria:

Subjects will be ineligible for this study based on any one of the following criteria:

1. With a chronic or acute disease that might interfere with the evaluation of Xolair therapy
2. Pregnancy or lactation
3. Current or prior malignancies (excluding non-melanoma skin carcinoma or carcinoma in situ of the cervix that has been adequately treated)
4. History of infection with human immunodeficiency virus (HSC-1), hepatitis B virus (HBV), or hepatitis C virus (HCV); or Hepatitis A virus (HAV)
5. Infections that require intravenous antibiotic therapy
6. Significant organ dysfunction, including cardiac, renal, liver, CNS, pulmonary, vascular, gastrointestinal, endocrine, or metabolic
7. Treatment with a humanized or chimeric antibody therapy within 4 weeks prior to study entry
8. Treatment with any investigational drugs or therapies within 2 weeks prior to study entry
9. Any use of oral, systemic corticosteroids within 2 weeks prior to study entry
10. Any use of topical agents for eczema or anti-pruritic agents 1 week prior to study entry.
11. Treatment with antihistamines within 4 days of the first skin test screen.
12. History of allergen immunotherapy within one year of the study start -

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2004-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nadeau, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Iyengar SR, Hoyte EG, Loza A, Bonaccorso S, Chiang D, Umetsu DT, Nadeau KC. Immunologic effects of omalizumab in children with severe refractory atopic dermatitis: a randomized, placebo-controlled clinical trial. Int Arch Allergy Immunol. 2013;162(1):89-93. doi: 10.1159/000350486. Epub 2013 Jun 27. PMID 23816920